CLINICAL TRIAL: NCT02564406
Title: Extracorporeal CO2 Removal in Hypercapnic Patients Who Failed Noninvasive Ventilation and Refuse Endotracheal Intubation: a Case Series
Brief Title: Extracorporeal CO2 Removal in Hypercapnic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Andrea Morelli, MD. Associate professor, University of Roma La Sapienza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3785
Record Dates: First submitted 2015-09-26; First posted 2015-09-30 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- hypercapnic patients (Experimental): patients with acute hypercapnic respiratory failure due to exacerbation of chronic obstructive pulmonary disease, refused endotracheal intubation after failing NIV and were treated withLow flow etracorporeal CO2 removal
  Interventions: Device: LOW FLOW EXTRACORPOREAL CO2 REMOVAL, PROLUNG ESTOR

INTERVENTIONS:
Device: LOW FLOW EXTRACORPOREAL CO2 REMOVAL, PROLUNG ESTOR

SUMMARY:
Noninvasive ventilation represents the standard of care for patients with exacerbation of chronic obstructive pulmonary disease. However, NIV fails in almost 30% of the most severe forms of acute hypercapnic respiratory failure and patients must undergo endotracheal intubation and invasive ventilation to restore adequate gas exchange. Under these circumstances, patients may express a clear intention not to be intubated.The aim of this study is to retrospectively assess efficacy and safety of noninvasive ventilation- plus-extracorporeal Co2 removal in patients who fail NIV and refuse endotracheal intubation.

DETAILED DESCRIPTION:
During a period of two years (from January 2013 to July 2015) 35 patients with acute hypercapnic respiratory failure due to exacerbation of chronic obstructive pulmonary disease, refused endotracheal intubation after failing NIV and were treated with extracorporeal Co2 removal plus NIV as last resort therapy.

The collected data of these patients will be retrospectively matched with data obtained from 35 historical controls who received conventional treatment with endotracheal intubation. The study will retrospectively compare intubation rate, acid base homeostasis, norepinephrine requirements (in the patients who due to clinical conditions were under norepinephrine before starting extracorporeal Co2 removal ) and coagulation parameters.

ELIGIBILITY:
Inclusion Criteria:

* exacerbation of chronic obstructive pulmonary disease
* failure of non invasive ventilation
* expression of a clear intention not to be intubated

Exclusion Criteria:

* alterations in mental status which do not allow to express a clear intention not to be intubated
* contraindications to anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
number of patients who avoided endotracheal intubation | 60 days

SECONDARY OUTCOMES:
Gas exchange homeostasis | 96 hrs
  pH, PaCO2, PaO2, bicarbonate, arterial lactate
Norepinephrine requirements | 30 days
  norepinephrine requirements in the patients who due to clinical conditions were under norepinephrine before starting the treatment with extracorporeal Co2 removal
coagulation | 30 days
  INR, pt, ptt. platelets
Day 28 mortality | 28 days
intra hospital mortality | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Morelli, MD, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Dept of Anesthesiology and Intensive Care, Rome, Italy

REFERENCES:
- [Background] Burki NK, Mani RK, Herth FJF, Schmidt W, Teschler H, Bonin F, Becker H, Randerath WJ, Stieglitz S, Hagmeyer L, Priegnitz C, Pfeifer M, Blaas SH, Putensen C, Theuerkauf N, Quintel M, Moerer O. A novel extracorporeal CO(2) removal system: results of a pilot study of hypercapnic respiratory failure in patients with COPD. Chest. 2013 Mar;143(3):678-686. doi: 10.1378/chest.12-0228. PMID 23460154
- [Background] Del Sorbo L, Pisani L, Filippini C, Fanelli V, Fasano L, Terragni P, Dell'Amore A, Urbino R, Mascia L, Evangelista A, Antro C, D'Amato R, Sucre MJ, Simonetti U, Persico P, Nava S, Ranieri VM. Extracorporeal Co2 removal in hypercapnic patients at risk of noninvasive ventilation failure: a matched cohort study with historical control. Crit Care Med. 2015 Jan;43(1):120-7. doi: 10.1097/CCM.0000000000000607. PMID 25230375